CLINICAL TRIAL: NCT00981162
Title: A Phase I/II Study of Sorafenib and Everolimus in Patients With Advanced Solid Tumors and Gemcitabine-Refractory Metastatic Pancreatic Cancer
Brief Title: Sorafenib Tosylate and Everolimus in Treating Patients With Advanced Solid Tumors and Metastatic Pancreatic Cancer That Does Not Respond to Gemcitabine Hydrochloride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 150109; NCI-2009-01326 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 150109 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IV Pancreatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Sorafenib; Everolimus; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (sorafenib tosylate and everolimus) (Experimental): Patients receive everolimus PO once daily and sorafenib tosylate PO twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Drug: everolimus; Other: laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study

INTERVENTIONS:
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Other: laboratory biomarker analysis — Correlative study
Other: pharmacogenomic studies — Correlative study
  Other Names: Pharmacogenomic Study
Other: pharmacological study — Correlative study
  Other Names: pharmacological studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of everolimus when given together with sorafenib tosylate and to see how well they work in treating patients with advanced solid tumors and metastatic pancreatic cancer that does not respond to gemcitabine hydrochloride. Sorafenib tosylate and everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib tosylate may also stop the growth of pancreatic cancer by blocking blood flow to the tumor. Giving sorafenib tosylate together with everolimus may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 6-month overall survival of patients with previously treated gemcitabine (gemcitabine hydrochloride)-refractory metastatic pancreatic cancer treated with the combination of sorafenib (sorafenib tosylate) and everolimus.

II. To determine the recommended Phase II dose of everolimus when administered in combination with sorafenib in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To determine the response rate, median survival, time to progression, CA 19.9 decline and toxicity spectrum of the combination in this patient population.

II. To characterize the pharmacokinetic (PK) profiles of sorafenib and everolimus when given in combination.

III. To explore the biomarkers that correlate with response to the study combination in patients previously treated with gemcitabine-refractory metastatic pancreas cancer.

OUTLINE: This is a phase I, dose-escalation study of everolimus, followed by a phase II study.

Patients receive everolimus (PO) once daily and sorafenib tosylate PO twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Phase I only: Histologically or cytologically confirmed solid tumors that are advanced and refractory to or lack life-prolonging treatments; patients with histologically or cytologically confirmed renal cell carcinoma and hepatocellular carcinoma will be eligible
* Phase II: Histologically or cytologically proven metastatic adenocarcinoma of pancreas that had progressed after one prior gemcitabine containing regimen, or progressed within 6 months of the completion of gemcitabine containing adjuvant regimen
* Patients must have measurable or assessable disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate hematological, renal and liver functions as determined by the following:
* Absolute neutrophil count (ANC) > 1500 cells/mm^3
* Hemoglobin >= 9g/dL
* Platelets >= 100,000 cells/mm^3
* Serum creatinine within institutional upper limit of normal (ULN) OR >= 60mll/min for patients with creatinine levels above institutional ULN
* Bilirubin =< 1.5 x ULN
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 times ULN (< 5 x ULN for patients with abnormal values attributable to liver metastases)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 times ULN (< 5 x ULN for patients with abnormal values attributable to liver metastases)
* International normalized ratio (INR) =< 1.5 (Anticoagulation is allowed if target INR =< 1.5 on a stable dose of warfarin or on a stable dose of low-molecular-weight (LMW) heparin for > 2 weeks at the first dose of study agent)
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L AND Fasting triglycerides =<2.5 x ULN; NOTE: in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Ability to understand and willingness to sign a written informed consent; a signed informed consent must be obtained prior to any study specific procedures
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation; men should use adequate birth control for at least three months after the last administration of sorafenib and everolimus

Exclusion Criteria:

* Phase II: Patients in whom histological or cryological diagnosis is not consistent with adenocarcinoma including adenosquamous, islet cell, cystoadenoma or cystadenocarcinoma, carcinoid, small or large cell carcinoma or lymphoma
* Phase II: Adenocarcinoma arising from a site other than the pancreas (distal bile duct, ampulla of vater or periampullary duodenum)
* Prior therapy with approved or investigational agents within 4 weeks prior to the start of treatment plan in this protocol
* Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN
* Any active infections
* Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA); patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management
* Cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event >= Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event >= CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known or suspected allergy to sorafenib, everolimus, other rapamycins (sirolimus, temsirolimus), their excipients, or any agent given in the course of this trial
* Any condition that impairs patient's ability to swallow whole pills
* Any malabsorption problem
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days of first study drug
* Urine protein:creatinine ratio >=1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of baseline
* Inability to comply with study and/or follow-up procedures
* History of concurrent malignancy or history of a second malignancy within the past 5 years
* Unable to provide informed consent
* Concomitant use of any medications or substances that are inhibitors or inducers of CYP3A enzyme, which include but not limited to phenytoin, carbamazepine, barbiturates, rifampin, Phenobarbital or St. Johns Wort
* Phase II: Prior treatment with mTOR inhibitors (e.g., sirolimus, temsirolimus, everolimus) or Ras-MAPK inhibitors (e.g., sorafenib)
* Any unresolved chronic toxicity greater than CTCAE grade 2 from previous anticancer therapy (except alopecia)
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent; topical or inhaled corticosteroids are allowed
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period; close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus (Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines)
* Severely impaired lung function as defined as spirometry and diffusing capacity of carbon monoxide (DLCO) that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air; patients are not required to undergo mandatory respiratory function tests at screening to be eligible unless medically necessary
* Severe and/or uncontrolled non-malignant liver disease such as cirrhosis or severe hepatic impairment defined as Child-Pugh class C
* A known history of human immunodeficiency virus (HIV) seropositivity
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods; if barrier contraceptives are being used, these must be continued throughout the trial by both sexes; hormonal contraceptives are not acceptable as a sole method of contraception
* Women of childbearing potential (WOCBP) that have a positive urine or serum pregnancy test within 7 days prior to the start of treatment
* Male patient whose sexual partner(s) are WOCBP who are not willing to use adequate contraception during the study and for 8 weeks after the end of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (Phase II) | Time from date of subject enrollment to the date of death due to any cause, assessed up to 6 months
  The estimated distribution of overall survival will be obtained using the product-limit based Kaplan-Meier method. Estimates of quantities such as median survival will be obtained.
Maximum tolerated dose of everolimus (Phase I) | 28 days
  Assessed by National Cancer Institute (NCI) CTCAE v3.0.

SECONDARY OUTCOMES:
Overall response rate (Phase II) | Up to 1 year
  Will be computed with a corresponding exact 95% confidence interval.
Differences in biomarkers between responders and non-responders (Phase II) | Baseline and days 1 and 15 of course 1
PK parameters (Phase II) | Baseline and days 1 and 15 of course 1
  Will be summarized in each cohort of patients. Comparison of PK parameters among the dose levels will be performed using non-parametric statistical methods for K-independent samples.
Correlation of predicted drug concentration or area under the curve (AUC) with biomarker response for each drug and/or in combination (Phase II) | Baseline and days 1 and 15 of course 1
Toxicity and adverse events as assessed by NCI CTCAE v3.0 | Up to 30 days post-treatment
  All toxicities and adverse events in the Phase I and Phase II portions will be summarized with frequencies and descriptive measures.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wee Ma, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - University of Colorado at Denver Health Sciences Center, Aurora, Colorado
  - Roswell Park Cancer Institute, Buffalo, New York